CLINICAL TRIAL: NCT03619343
Title: A New Treatment Modality for the Postoperative Muscular Pain Management in Pylorus Preserving Pancreaticoduodenectomy: a Double-blind Randomized Control Trial
Brief Title: Postoperative Muscular Pain, ETOIMS (Electrical Twitch Obstructive Intramuscular Stimulation)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Joon Seong Park, Professor,, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2018-0100
Record Dates: First submitted 2018-07-27; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Disease Status of Pancreatobiliary Tract , ( Especially Who Need to Undergo Pancreaticoduodenectomy)

STUDY DESIGN:
Intervention Model Description: Control Intervention : ETOIMS apply group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No ETOIMS arm (Experimental): When the abdominal wound is closed, the operator performs needle insertion at 14 sites near the incision site under the guidance of ultrasonography.
  Interventions: Procedure: ETOIMS(Electrical Twitch Obtaining Intramuscular Stimulation)
- ETOIMS arm (Active Comparator): When the abdominal wound is closed, the operator performs needle insertion at 14 sites near the incision site under the guidance of ultrasonography. When the needle is in the abdominal muscle, the operator performs muscle stimulation for about 10 seconds per needle insertion.
  Interventions: Procedure: ETOIMS(Electrical Twitch Obtaining Intramuscular Stimulation)

INTERVENTIONS:
Procedure: ETOIMS(Electrical Twitch Obtaining Intramuscular Stimulation) — When the abdominal wound is closed, the operator performs needle insertion at 14 sites near the incision site under the guidance of ultrasonography. When the needle is in the abdominal muscle, the operator performs muscle stimulation for about 10 seconds per needle insertion.

SUMMARY:
Pancreaticoduodenectomy is inevitably an operation requiring extensive skin and muscle incision, resulting in postoperative pain resulting in limitation of the patient's early exercise and function. ETOIMS(Electrical Twitch Obstructive Intramuscular Stimulation) is used to relieve muscle pain and relax muscles. ETOIMS is a method to relieve pain by stimulating muscle in myofascial pain syndrome. ETOIMS as an effective new treatment for pain after pylorus preserving pancreaticoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pancreatoduodenectomy in Gangnam Severance Hospital, Seoul, Korea
* Patients who are able to perform daily activities before surgery and were able to walk independently.
* Adults over 20

Exclusion Criteria:

* Patients with history of previous open surgery

  * Patients who are not able to exercise due to severe musculoskeletal pain except surgery-related diseases
  * Patients who can not walk because of difficulty breathing related to myalgia
  * Patients who can not exercise due to severe musculoskeletal pain
  * Patients who had a limb defect before surgery and were unable to walk without assistive devices and others
  * Pregnant / lactating mothers
  * Patients who have cognitive impairment and can not answer the questionnaire
  * Patients with Pacemaker
  * Patients who can not read the consent form

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-02-18 (Estimated); Study Completion 2019-06-18 (Estimated)

PRIMARY OUTCOMES:
Pain: VAS (visual analogue scale) | AM 7:00 morning at Preoperative day and the day following surgery before discharge (Postoperative day 1 - Postoperative day 10)
  The primary outcome of this study was the postoperative pain score (VAS score) in patients undergoing ETOIMS during surgery. The type of surgery in the experimental group and the control group is the same and the same analgesic agent (IV PCA, Wound PCA) is used. The pain score is measured at 7 o'clock every morning from the day following surgery to discharge (about Postoperative day 10) to confirm the reduced pattern.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park J, Kim HS, Park JH, Park YG, Shin S, Park JE, Hwang S, Jun SY, Park JS. Effectiveness of Intramuscular Electrical Stimulation on Postsurgical Nociceptive Pain for Patients Undergoing Open Pancreaticoduodenectomy: A Randomized Clinical Trial. J Am Coll Surg. 2020 Sep;231(3):339-350. doi: 10.1016/j.jamcollsurg.2020.06.008. Epub 2020 Jul 2. PMID 32623088